CLINICAL TRIAL: NCT01845480
Title: The Wildcat Wellness Coaching Trial: Home-based Obesity Prevention and Health Promotion in Children and Adolescents
Brief Title: The Wildcat Wellness Coaching Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Richard R. Rosenkranz, Associate Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KSU-CHE-SRO-WWCT
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Health Promotion and Obesity Prevention
Keywords: health promotion; obesity prevention; Childhood obesity; home-based; Lifestyle intervention; Body composition; quality of life; physical activity; nutrition
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthful eating phys activity coaching (Experimental): The healthful eating and physical activity skills coaching intervention is designed to help children set goals and self-monitor healthful eating and physical activity; teach kitchen skills for fruit and vegetable snack preparation; teach children enjoyable physical activities to do at home (e.g., dancing); and provide modeling and social support for physical activity and healthful eating.
  Interventions: Behavioral: Wellness coaching
- Health education coaching (Active Comparator): Health education coaching is designed to help children set goals and self-monitor behavior; educate children on a range of relevant health promotion behaviors (e.g., tooth brushing, not smoking, physical activity, etc.); and provide modeling and social support for practicing healthful behavior.
  Interventions: Behavioral: Wellness coaching

INTERVENTIONS:
Behavioral: Wellness coaching — Wellness coaching that includes modeling, goal setting, self-monitoring, social support, and health behavior education
  Other Names: health coaching

SUMMARY:
Female children (aged 8-13 years) will be recruited through posted flyers, newspaper ads, and word of mouth in the Manhattan, KS area. After laboratory assessment, recruited participants will be randomly assigned to either healthful eating and physical activity skills coaching or general health education coaching intervention conditions. For both conditions, research assistants will serve as wellness coaches and deliver 12 intervention sessions in the home of each participating child.

Assessments will be completed at baseline, intervention end (3 months), and follow-up (6 months), comprising biomedical and psychosocial measures. Biomedical measurements to be obtained include:

* body composition (DEXA, tetrapolar bioimpedance, body mass index, waist circumference)
* blood pressure (automated sphygmomanometer),
* pulmonary function tests (forced expiratory flow in 1-sec, forced vital capacity, forced expiratory flow at 25-75% of vital capacity),
* unstimulated whole (mixed) saliva passive drool to detect markers of inflammation,
* and physical activity levels (7-day accelerometry).

Psychosocial measurements include:

* fruit and vegetable consumption (Child Dietary Questionnaire)
* self efficacy,
* enjoyment
* quality of life (Peds QL).

Inclusion criteria are:

* being female
* aged 8-13 years
* with parental consent,
* residing within a 40-minute drive
* being available for 12 home coaching visits and three lab assessments.

Exclusion criteria are

* having developmental delay or psychiatric problems,
* any illness, injury, condition, or disease that would prevent participation in moderate-to-vigorous physical activity,
* taking weight-altering medications
* participating in any other health behavior change program.

The objectives of this study are to determine

* whether both types of the home-based coaching interventions are feasible
* whether the healthful eating and physical activity skills coaching intervention is more efficacious, relative to the general health education coaching group, in preventing increases in body fat percentage, body mass index percentile, waist circumference, systolic and diastolic blood pressure, and sedentary behavior
* whether the healthful eating and physical activity skills coaching intervention is more efficacious, relative to the general health education coaching group, in facilitating increases in quality of life, moderate-to-vigorous physical activity, enjoyment of physical activity and fruit and vegetable consumption, and self-efficacy for physical activity and fruit and vegetable consumption.

We hypothesize that the research project will be successful in recruiting and retaining participating families, training research assistants to deliver the intervention components, and that both of the coaching conditions will be well received and appreciated by participating families. We hypothesize that the healthful eating and physical activity skills coaching intervention will be more effective than the support coaching condition in preventing increases in blood pressure, airway dysfunction and adiposity. We expect that both intervention conditions will show improvements to pediatric quality of life measures, but that the healthful eating and physical activity skills coaching intervention will be more effective than general health education coaching condition in increasing physical activity, physical activity enjoyment and self efficacy, fruit and vegetable consumption, and fruit and vegetable enjoyment and self-efficacy.

DETAILED DESCRIPTION:
Obesity is associated with increased chronic disease risk, and therefore poses a major public health problem (Lobstein et al., 2004). In 2011, the Centers for Disease Control and Prevention estimated that obesity affects about 12.5 million children and teens, or 17% of the US population. This is a marked increase from the ~5% rate of obesity found in this population in the late 1960s. Barlow (2007) points out that the complexity of obesity prevention lies less in the identification of target health behaviors, and much more in a process of influencing families to change behaviors when habits, culture, and environment promote less physical activity and more energy intake.

Obesity prevention interventions may not be effective or sustainable without impacting home environments (Rosenkranz & Dzewaltowski, 2008). Conwell et al. (2010) suggest that home-based programs may offer significant advantages over center-based programs by offering better accessibility and convenience. Wellness coaching has shown promise for improving health behaviors related to chronic disease (Lawn & Schoo, 2010), but no published study has used a wellness coaching childhood obesity prevention model in the home environment.

The primary aim of this trial is to determine whether the home-based wellness coaching delivery model is feasible as an obesity prevention intervention strategy in the community setting. The secondary objective is to determine the comparative effectiveness of the two wellness coaching interventions.

Female children (aged 8-13 years) will be recruited through posted flyers, newspaper ads, and word of mouth in the Manhattan, KS area. After laboratory assessment, recruited participants will be randomly assigned to either healthful eating and physical activity skills coaching or general health education coaching intervention conditions. For both conditions, research assistants will serve as wellness coaches and deliver 12 intervention sessions in the home of each participating child. Assessments will be completed at baseline, intervention end (3 months), and follow-up (6 months), comprising biomedical and psychosocial measures.

We hypothesize that the research project will be successful in recruiting and retaining participating families, training research assistants to deliver the intervention components, and that both of the coaching conditions will be well received and appreciated by participating families. We hypothesize that the healthful eating and physical activity skills coaching intervention will be more effective than the support coaching condition in preventing increases in blood pressure, airway dysfunction and adiposity. We expect that both intervention conditions will show improvements to pediatric quality of life measures, but that the healthful eating and physical activity skills coaching intervention will be more effective than general health education coaching condition in increasing physical activity, physical activity enjoyment and self efficacy, fruit and vegetable consumption, and fruit and vegetable enjoyment and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Being a female aged 8 to 13 years with consenting parent or guardian
* Family willing to participate in home-based behavioral intervention

Exclusion Criteria:

* Having developmental delay or psychiatric problems.
* Having any illness, injury, condition, or disease that would prevent participation in moderate-to-vigorous physical activity.
* Not living within 40 miles of Kansas State University campus in Manhattan, KS.
* Taking weight-altering medications, or participating in any other weight control program.

Ages: 8 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2017-09-20 (Estimated); Study Completion 2017-10-13 (Estimated)

PRIMARY OUTCOMES:
body mass index Z-score | change from baseline BMIz at 6 months
  CDC age- and sex-referenced body mass index standardized score

SECONDARY OUTCOMES:
Quality of life | change from baseline at 6 months
  Quality of life (PedsQL scales of physical functioning, social functioning, school functioning, emotional functioning)

OTHER OUTCOMES:
Consumption of fruits and vegetables | change from baseline at 6 months
  Daily consumption of fruits and vegetables
Physical activity | change from baseline at 6 months
  Weekly step count, minutes per day of moderate-to-vigorous physical activity, minutes per day of sedentary behavior
body fat percentage | change from baseline at 6 months
  DEXA-assessed body fat percentage
Waist circumference | change from baseline at 6 months
  Gulick tape measured horizontal distance around waist during exhale at midpoint of rib and iliac crest

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Rosenkranz, Rosenkranz, Principal Investigator — Kansas State University
Locations (1):
- Physical Activity & Nutrition Clinical Research Consortium, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cull BJ, Rosenkranz SK, Dzewaltowski DA, Teeman CS, Knutson CK, Rosenkranz RR. Wildcat wellness coaching feasibility trial: protocol for home-based health behavior mentoring in girls. Pilot Feasibility Stud. 2016 Jun 1;2:26. doi: 10.1186/s40814-016-0066-y. eCollection 2016. PMID 27965845
- See also: Published protocol paper — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-016-0066-y